CLINICAL TRIAL: NCT02048722
Title: Multicenter, Open-Label Phase II Study of Daily Oral Regorafenib for Chemotherapy-Refractory, Metastatic and Locally Advanced Angiosarcoma
Brief Title: Daily Oral Regorafenib for Chemotherapy-Refractory, Metastatic and Locally Advanced Angiosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Bayer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 13S02; NCI-2013-02278 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00087654 (Other: Northwestern University IRB#); ONC-2013-129; NU 13S02 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-01-29 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Adult Angiosarcoma; Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Hemangiosarcoma; Sarcoma | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (regorafenib) (Experimental): Patients receive regorafenib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — Given PO
  Other Names: BAY 73-4506; multikinase inhibitor BAY 73-4506; Stivarga

SUMMARY:
The purpose of this study is to see whether a drug called regorafenib might be effective in treating angiosarcoma. This study is for patients who have angiosarcoma that has gotten worse after they received chemotherapy. Regorafenib is a type of drug called a kinase inhibitor. Regorafenib interferes with how some kinase proteins work. Some of these kinases in cancer cells might normally help the cancer cells grow or form new blood vessels that could feed a growing tumor. By blocking these proteins, regorafenib may help stop the growth of certain cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the progression-free survival (PFS) at 4 months with daily oral regorafenib (160 mg) in previously treated locally advanced/metastatic angiosarcoma patients

SECONDARY OBJECTIVES:

I. Progression-free rate at 3 and 6 months. II. Progression-free survival. III. Overall survival (up to 5 years). IV. Response rate (by Response Evaluation Criteria in Solid Tumors [RECIST] version [v] 1.1).

V. Rate and duration of tumor control (complete response [CR] + partial response [PR] + stable disease [SD]).

VI. Safety/tolerability of regorafenib.

OUTLINE:

Patients receive regorafenib orally (PO) once daily (QD) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 4 months
* Histologically confirmed angiosarcoma
* Tumor deemed unresectable or metastatic
* Measurable disease per RECIST v 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Progressive disease under last palliative therapy with a history of prior ifosfamide, doxorubicin or taxane therapy for angiosarcoma; up to 4 prior therapies are allowed
* All acute toxic effects of any prior treatment have resolved to grade 1 or less (by National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v 4.0) at the time of registration; NOTE: Exceptions to this criterion will include alopecia and fatigue
* Total bilirubin =< 1.5 x the upper limits of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Alkaline phosphatase limit =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Lipase =< 1.5 x the ULN
* Serum creatinine =< 1.5 x the ULN
* International normalized ratio (INR)/partial thromboplastin time (PTT) < 1.5 x ULN
* Platelet count > 100000/mm^3
* Hemoglobin > 9 g/dL
* Absolute neutrophil count > 1500/mm^3
* If baseline urine protein creatinine (UPC) >= 1, a 24-hour urine protein must be assessed; patients must have a 24-hour urine protein value < grade 3 (> 3.5 g/24 hours) to be eligible
* NOTE: Blood transfusion to meet the above criteria will not be allowed; NOTE: Patients who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists; close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug; post-menopausal women (defined as age >= 50 years and no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at registration until at least 3 months after the last dose of study drug; the definition of adequate contraception will be based on the judgment of the principal investigator
* Subject must be able to swallow and retain oral medication
* Subjects must be able to understand and be willing to sign the written informed consent form; a signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure

Exclusion Criteria:

* Uncontrolled hypertension (systolic pressure > 140 mmHg or diastolic pressure > 90 mmHg on repeated measurement) despite optimal medical management
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association > class II
  * Active coronary artery disease
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before registration, or myocardial infarction within 6 months before registration
* Evidence or history of bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding event grade 3 within 4 weeks prior to registration
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months of informed consent
* Subjects with any previously untreated or concurrent cancer unrelated to angiosarcoma; NOTE: Exceptions include cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor; subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before registration are allowed; all treatments must have been completed at least 3 years prior to registration
* Patients with pheochromocytoma
* Patients with severe hepatic impairment (Child-Pugh class C)
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Ongoing infection > grade 2
* Evidence of significant central nervous system disease including seizure disorder requiring medication, symptomatic metastatic brain or meningeal tumors
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Renal failure requiring hemo-or peritoneal dialysis
* Dehydration > grade 1
* Interstitial lung disease with ongoing signs and symptoms at the time of registration
* Pleural effusion or ascites that causes respiratory compromise (>= grade 2 dyspnea)
* History of organ allograft (including corneal transplant)
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
* Any malabsorption condition
* Evidence of abdominal fistula, gastrointestinal (GI) perforation or intraabdominal abscess
* Women who are pregnant or breast-feeding
* Concurrent anti-cancer therapy (chemotherapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than study treatment (regorafenib)
* Prior use of regorafenib
* Prior use of sorafenib
* Use of cytotoxic chemotherapy within 21 days of registration
* Use of targeted therapy within two half-lives of registration
* Radiation directed at target lesion within 28 days of registration
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before registration
* Therapeutic anticoagulation with Vitamin-K antagonists (e.g., warfarin) or with heparins and heparinoids; NOTE: Prophylactic anticoagulation as described below is allowed:

  * Low dose warfarin (1 mg orally, once daily) with prothrombin time (PT)-international normalized ratio (INR) =< 1.5 x ULN is permitted; infrequent bleeding or elevations in PT-INR have been reported in some subjects taking warfarin while on regorafenib therapy; therefore, subjects taking concomitant warfarin should be monitored regularly for changes in PT, PT-INR or clinical bleeding episodes
  * Low dose aspirin (=< 100 mg daily)
  * Prophylactic doses of heparin
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Agulnik, M.D., Principal Investigator — Northwestern University
Locations (7):
- United States (7):
  - Sarcoma Oncology Center, Santa Monica, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University-St. Louis, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened for enrollment March 12, 2014 with the first patient starting treatment June 13, 2014. A total of 31 patients were treated under the protocol. The study was permanently suspended to further enrollment August 5, 2019.
Period: 2 Cycles of Treatment
Arm/Group | Treatment (Regorafenib)
Started | 31
Attempted 1st Cycle | 31
Attempted 2nd Cycle | 23
Completed | 23
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 4
Not completed — Progressive Disease | 2
Period: Reached 1st Response/Continued Treatment
Arm/Group | Treatment (Regorafenib)
Started | 23
Assessed for First Response | 23
Went on to Cycle 3 and Beyond | 13
Completed | 13
Not Completed | 10
Not completed — Progressive Disease | 10
Period: Follow up 5 Years or Cut of Timepoint
Arm/Group | Treatment (Regorafenib)
Started (All patients that have one does of study drug go into follow up after discontinuing treatment. Patients followed for 5 years or until October 12, 2021, whichever comes first.) | 31
Completed | 4
Not Completed | 27
Not completed — Death | 24
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: This includes patients that started study treatment. Any patients who signed consent but never initiated treatment (screenfails) are not included.
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 31
Age, Customized [Mean (Standard Deviation); unit: years] | 64.32 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 31
Type of disease [Count of Participants; unit: Participants]
  Metastatic | 21
  Locally advanced/Unresectable | 9
  Not reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at 4 Months
Description: The progression-free survival (PFS) at 4 months will be defined as the number of patients with progression absent at 4 months divided by the total number of evaluable study patients. This will be measured from start of treatment until time of progression or death, whichever occurs first and will be estimated using Kaplan-Meier methods and reported as a survival probability.
  Progression will be evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in RECIST v 1.1. Progression will be defined as:
  Progressive disease (PD): > 20% increase in the sum diameters of target lesions, taking as reference the smallest sum diameters while on study. The sum diameters must also demonstrate an absolute increase of 5 mm. The appearance of one or more new lesions also qualifies as PD.
Time Frame: At 4 months (of treatment)
Population: 8 Patients were not included due to the following reasons: progressive disease, patient refused further treatment (withdrawal of consent for further treatment), toxicity. This was due to data having either missing time points or "cycle 1" or "Cycle 1: follow up" missing from the dataset at the time of the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients alive
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 23
percentage of patients alive | 52.17 [35.28 to 77.16]

2. Secondary Outcome: Progression-Free Survival (PFS) at 3 and 6 Months
Description: The progression-free survival (PFS) at 3 and 6 months will be defined as the number of patients with progression absent at 3 months and 6 months divided by the total number of evaluable study patients. This will be measured from start of treatment until time of progression or death, whichever occurs first and will be estimated using Kaplan-Meier methods and reported as a survival probability.
  Progression will be evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in RECIST v 1.1. Progression will be defined as:
  Progressive disease (PD): > 20% increase in the sum diameters of target lesions, taking as reference the smallest sum diameters while on study. The sum diameters must also demonstrate an absolute increase of 5 mm. The appearance of one or more new lesions also qualifies as PD.
Time Frame: Assessed at 3 months and 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage patients alive
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 23
percentage patients alive
  3 months | 56.52 [39.5 to 80.89]
  6 months | 47.83 [31.21 to 73.29]

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: The median progression-free rate (PFR) will be defined as the number of patients with progression absent divided by the total number of evaluable study patients. This will be measured from start of treatment until time of progression or death, whichever occurs first for up to 5 years and will be estimated using Kaplan-Meier methods.
  Progression will be evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in RECIST v 1.1. Progression will be defined as:
  Progressive disease (PD): > 20% increase in the sum diameters of target lesions, taking as reference the smallest sum diameters while on study. The sum diameters must also demonstrate an absolute increase of 5 mm. The appearance of one or more new lesions also qualifies as PD.
Time Frame: The duration of time from start of treatment until time of progression, up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 23
months | 5.49 [1.84 to 9.53]

4. Secondary Outcome: Overall Survival
Description: Overall survival will be defined as the time from start of treatment until death from any cause and will be estimated using Kaplan-Meier methods and reported as a survival probability. Patients that are alive at the time of data analysis will be censored at the date of known survival status.
Time Frame: From start of treatment up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 23
months | 14.06 [9.76 to 22.24]

5. Secondary Outcome: Response Rate
Description: Imaging (such as a CT scan) will be done at baseline (within 4 weeks before the first dose) then after every 2 cycles while on treatment for tumor response evaluation. Response will be evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in RECIST v 1.1. Best response of each patient will be used and responses will be defined as the following:
  Complete response (CR): Disappearance of all target lesions Partial response (PR): > 30% decrease in the baseline sum diameters of target lesions
Time Frame: At baseline and after every 2 cycles, up to 12 cycles where one cycle is 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 23
participants
  Complete Response | 2
  Partial Response | 2

6. Secondary Outcome: Rate of Tumor Control
Description: Imaging will be used at baseline then after every 2 cycles while on treatment to measure tumor size and response to treatment, the data collected from all patients on study will be used to calculate the rate and duration of tumor control.
  Response will be evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in RECIST v 1.1. Response and stable disease will be defined as the following:
  Complete response (CR): Disappearance of all target lesions Partial response (PR): > 30% decrease in the baseline sum diameters of target lesions Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: At baseline and after every 2 cycles, up to 12 cycles where one cycle is 28 days
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 23
patients
  Complete Response | 2
  Partial Response | 2
  Stable Disease | 9

7. Secondary Outcome: Number of Grade 1, 2, 3, 4, and 5 Related Adverse Events Observed During Study Treatment (Defined by CTCAE v 4.0)
Description: Overall worst grade related toxicity (number of patients) was collected from the start of treatment until 30 days post the last treatment where patients were treated until progressive disease or unacceptable toxicity or patient withdrawal of treatment. All Adverse events that were determined to be at least possibly related to treatment are reported.
  All adverse events will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  The severity of an AE is graded as follows:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities.
  Moderate (grade 2): the event causes discomfort that affects normal daily activities.
  Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status.
  Life-threatening (grade 4): the patient was at risk of death at the time of the event.
  Fatal (grade 5): the event caused death
Time Frame: From treatment initiation though 30 days post the last treatment for a max of 12 cycles where one cycle is 28 days
Population: At the time of data pull (12/02/2019) for this outcome measure two patients remained on treatment. Any subsequent AEs determined to be related to treatment for these patients is not included here.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Regorafenib)
Number analyzed (Participants) | 31
Participants
  Blood and lymphatic system disorders: Grade 1 | 5
  Blood and lymphatic system disorders: Grade 2 | 3
  Blood and lymphatic system disorders: Grade 3 | 3
  Blood and lymphatic system disorders: Grade 4 | 0
  Blood and lymphatic system disorders: Number of patients who didn't experience any grade | 20
  Endocrine disorders: Grade 1 | 1
  Endocrine disorders: Grade 2 | 0
  Endocrine disorders: Grade 3 | 0
  Endocrine disorders: Grade 4 | 0
  Endocrine disorders: Number of patients who didn't experience any grade | 30
  Eye disorders: Grade 1 | 2
  Eye disorders: Grade 2 | 0
  Eye disorders: Grade 3 | 0
  Eye disorders: Grade 4 | 0
  Eye disorders: Number of patients who didn't experience any grade | 29
  Gastrointestinal disorders: Grade 1 | 14
  Gastrointestinal disorders: Grade 2 | 9
  Gastrointestinal disorders: Grade 3 | 3
  Gastrointestinal disorders: Grade 4 | 0
  Gastrointestinal disorders: Number of patients who didn't experience any grade | 5
  General disorders: Grade 1 | 11
  General disorders: Grade 2 | 8
  General disorders: Grade 3 | 4
  General disorders: Grade 4 | 0
  General disorders: Number of patients who didn't experience any grade | 8
  Infections and infestations: Grade 1 | 1
  Infections and infestations: Grade 2 | 2
  Infections and infestations: Grade 3 | 0
  Infections and infestations: Grade 4 | 0
  Infections and infestations: Number of patients who didn't experience any grade | 28
  Injury, poisoning and procedural complications: Grade 1 | 0
  Injury, poisoning and procedural complications: Grade 2 | 1
  Injury, poisoning and procedural complications: Grade 3 | 0
  Injury, poisoning and procedural complications: Grade 4 | 0
  Injury, poisoning and procedural complications: Number of patients who didn't experience any grade | 30
  Metabolism and nutrition disorders: Grade 1 | 10
  Metabolism and nutrition disorders: Grade 2 | 4
  Metabolism and nutrition disorders: Grade 3 | 5
  Metabolism and nutrition disorders: Grade 4 | 0
  Metabolism and nutrition disorders: Number of patients who didn't experience any grade | 12
  Investigations: Grade 1 | 14
  Investigations: Grade 2 | 2
  Investigations: Grade 3 | 3
  Investigations: Grade 4 | 1
  Investigations: Number of patients who didn't experience any grade | 11
  musculoskeletal and connective tissue disorders: Grade 1 | 7
  musculoskeletal and connective tissue disorders: Grade 2 | 3
  musculoskeletal and connective tissue disorders: Grade 3 | 1
  musculoskeletal and connective tissue disorders: Grade 4 | 0
  musculoskeletal and connective tissue disorders: Number of patients who didn't experience any grade | 20
  Neoplasms benign, malignant and unspecified: Grade 1 | 1
  Neoplasms benign, malignant and unspecified: Grade 2 | 0
  Neoplasms benign, malignant and unspecified: Grade 3 | 0
  Neoplasms benign, malignant and unspecified: Grade 4 | 0
  Neoplasms benign, malignant and unspecified: Number of patients who didn't experience any grade | 30
  Nervous system disorders: Grade 1 | 11
  Nervous system disorders: Grade 2 | 2
  Nervous system disorders: Grade 3 | 1
  Nervous system disorders: Grade 4 | 0
  Nervous system disorders: Number of patients who didn't experience any grade | 17
  Psychiatric disorders: Grade 1 | 3
  Psychiatric disorders: Grade 2 | 1
  Psychiatric disorders: Grade 3 | 2
  Psychiatric disorders: Grade 4 | 0
  Psychiatric disorders: Number of patients who didn't experience any grade | 25
  Renal and urinary disorders: Grade 1 | 0
  Renal and urinary disorders: Grade 2 | 1
  Renal and urinary disorders: Grade 3 | 0
  Renal and urinary disorders: Grade 4 | 0
  Renal and urinary disorders: Number of patients who didn't experience any grade | 30
  Respiratory, thoracic and mediastinal disorders: Grade 1 | 9
  Respiratory, thoracic and mediastinal disorders: Grade 2 | 1
  Respiratory, thoracic and mediastinal disorders: Grade 3 | 1
  Respiratory, thoracic and mediastinal disorders: Grade 4 | 0
  Respiratory, thoracic and mediastinal disorders: Number of patients who didn't experience any grade | 20
  Skin and subcutaneous tissue disorders: Grade 1 | 14
  Skin and subcutaneous tissue disorders: Grade 2 | 6
  Skin and subcutaneous tissue disorders: Grade 3 | 1
  Skin and subcutaneous tissue disorders: Grade 4 | 0
  Skin and subcutaneous tissue disorders: Number of patients who didn't experience any grade | 10
  Vascular disorders: Grade 1 | 3
  Vascular disorders: Grade 2 | 8
  Vascular disorders: Grade 3 | 4
  Vascular disorders: Grade 4 | 0
  Vascular disorders: Number of patients who didn't experience any grade | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each patient from the initiation of treatment up until 30 days post last dose of treatment for a maximum of 12 cycles for any patient (where 1 Cycle = 28 days).
Description: Due to data collection methods, some serious adverse event (SAEs) data maybe captured within the other adverse event data information. There are patients currently on treatment and these sections will be updated with complete information at the study completion. SAEs for any patients that were screenfails (i.e., signed consent but never started study treatment) have been removed from these results. These patients were not included in the participant flow and baseline characteristics section.
Arm/Group | Treatment (Regorafenib)
All-Cause Mortality (participants affected / at risk) | 24/31
Serious Adverse Events (participants affected / at risk) | 15/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Regorafenib) (N=31)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient experienced chest pain at the time of the event
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient experienced acute kidney injury, anemia and hyperkalemia at the time of the event.
Intractable pain (General disorders) | 1 (1)
Vascular Disorder (Vascular disorders) | 1 (1) — Patient experienced dizziness at the time of this event.
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) — Patient experienced retroperitoneal hemorrhage at the time of this event.
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) — Patient with ileus and Takutsubo cardiomyopathy at the time of the event.
Nausea (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Generalized weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient experienced confusion at the time of the event.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient also experienced a thromboembolic event and hematuria at the time of this event.
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neck pain (General disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) — Patient also with anorexia at the time of the event
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient also experienced cough during this event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Regorafenib) (N=31)
Anemia (Blood and lymphatic system disorders) | 14
Leukocytosis (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 16
Oral dysesthesia (Gastrointestinal disorders) | 3
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 11
Chills (General disorders) | 2
Edema face (General disorders) | 2
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 23
Fever (General disorders) | 6
Gait disturbance (General disorders) | 5
General disorders and administration site conditions - Other, specify (General disorders) | 2
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 8
Gum infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Peripheral nerve infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 3
Hip fracture (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 9
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 7
INR increased (Investigations) | 5
Investigations - Other, specify (Investigations) | 2
Lipase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 16
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 11
Serum amylase increased (Investigations) | 1
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Trismus (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Ataxia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 9
Movements involuntary (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 6
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 8
Acute kidney injury (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 9
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 17
Hypotension (Vascular disorders) | 4
Vascular disorders - Other, specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT02048722/Prot_SAP_000.pdf